CLINICAL TRIAL: NCT04659668
Title: An Open-Label Uncontrolled Single Centre Study for the Evaluation of the Performance Characteristics (Efficacy and Safety) of the Dermal Filler MMG-23-04-2019 (Hyaluronic Acid 2,0%) for Female Intimate Area Hydration and Atrophy of the Vagina.
Brief Title: Evaluation of the Efficacy and Safety of the Dermal Filler for Female Intimate Area Hydration and Atrophy of the Vagina.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD/MMG-23-04-2019
Record Dates: First submitted 2020-11-20; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Vaginal Atrophy; Vulvovaginal Signs and Symptoms; Dyspareunia; Urinary Incontinence
MeSH Terms: conditions — Dyspareunia; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MMG-23-04-2019 (Experimental): MMG-23-04-2019 is composed by sodium hyaluronate at concentration of 2% (20 mg/ml) with 1,4-Butanediol diglycidyl ether (BDDE) acting as a cross-linking agent, in aqueous solution at physiological pH. The filler of 1ml is administered once or twice depending on the individual necessity.
  Interventions: Device: MMG-23-04-2019

INTERVENTIONS:
Device: MMG-23-04-2019 — The dermal filler MMG-23-04-2019 is applied to the female intimate area (intramucosal administration) of vaginal vestibule, vaginal walls, clitoris, "G" spot.

SUMMARY:
The study is an open-label uncontrolled single-center study for the evaluation of the Performance characteristics (efficacy and safety) of the dermal filler "MMG-23-04-2019" on the female genital area for the medicinal, functional and reconstructive indications.

DETAILED DESCRIPTION:
The Dermal Filler is recommended for the female intimate areas, especially the internal area of the vagina (vaginal vestibule, introitus, vaginal walls, clitoris, "G" spot) for the following indications: vaginal dryness or discomfort, vaginal atrophy.

The main functional ingredient is cross-linked hyaluronic acid of non-animal origin, produced through bacterial fermentation.

The MMG-23-04-2019 is contained in pre-filled, graduated and disposable sterile syringe with Luer Lock adapter with 1 ml of net content and 20 mg/ml hyaluronic acid.

The MMG-23-04-2019 has been classified as a Class III medical device under Annex IX of Directive MDD 93/42 EEC since it is a long-term, invasive and absorbable medical device.

ELIGIBILITY:
Inclusion Criteria:

* Female subject aged ≥18;
* Subject presenting vaginal atrophy, dryness, dyspareunia or discomfort in the intimate area;
* Subject who presents no other type of pathology of the area to be treated;
* Subject who is willing to abstain from any cosmetic or surgical procedures in the treatment area during the clinical investigation;
* Subject who is willing to participate in all study related activities and who is available for the duration of their participation in the investigation for follow-up;
* Absence of a history of significant hypersensitivity to food and drugs or known sensitivity to hyaluronic acid;
* Clinically and anamnestic healthy individual;
* Arterial blood pressure (BP) (after 5 min. at rest in the supine position) systolic 90 - 140 mmHg and diastolic 50 - 90 mmHg;
* Heart rate (HR) (after 5 min. at rest in the supine position) over 50 beats/min and less than 90 beats/min;
* Respiratory rate between 12 - 24 breaths/min;
* An axillar body temperature of up to 37 degrees celsius;
* Clinical-laboratory examinations within the reference ranges or with no clinically significant abnormalities;
* Negative AIDS/HIV test;
* Negative pregnancy test for the women with reproductive potential;
* A reliable and acceptable method of contraception for the women of child-bearing potential:
* Signed written Informed Consent Form

Exclusion Criteria:

* Subject with known sensitivity to hyaluronic acid or significant hypersensitivity to food and drugs;
* Subject with a history of vulvar cancer and/or previous regional radiotherapy;
* Subject with genital prolapse with a surgical indication or stress incontinence with a surgical indication;
* A subject who suffers from vaginism;
* Subject with genital bleeding of unknown origin;
* Subject with frequent or present active herpes simplex or herpes zoster local infection or active herpes simplex or herpes zoster infection in other sites;
* Subject with a history of frequent or active local dermatitis (of the injection site), vulvar scaly papilloma, mycosis; bacterial infection or laboratory tests indicating for such;
* A subject suffering from autoimmune diseases or who are undergoing treatment with immunosuppressors or immunotherapy;
* Subject with uncontrolled systemic diseases or who are undergoing current treatment with antihypertensives, steroid anti-inflammatory drugs anticoagulants, aspirin, major antidepressants;
* Pregnancy, postpartum period (6 months), lactation or post-lactation period (6 months);
* Absence of a reliable and effective method of contraception for a subject with childbearing potential;
* Subjects who are currently receiving another investigational treatment or who had participated in another clinical investigation within 30 days prior to study enrollment;
* A subject who suffer from another medical condition or who are receiving medication that in the Principal Investigator's judgment would prohibit the inclusion in the study;
* Subject with limited mental activity and consistent comprehension ability; sportsmen and individuals on strenuous physical loading; prisoners;
* Refusal to sign the Informed Consent Form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender-based pathology.
Enrollment: 37 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Vaginal Maturation Index (VMI) absolute change | From baseline to Day 60 (up to 8 weeks).
  Improvement in the properties of the vaginal wall, measured by the VMI.
Treatment-Emergent Adverse Events [Safety and Tolerability] | From screening through study completion, an average of 60 days - daily.
  Frequency and severity of adverse events (AEs) and adverse device effect

SECONDARY OUTCOMES:
The change in the Gloria Bachmann Vaginal Health Index (VHI) | From baseline to Day 30 (4 weeks) and Day 60 (up to 8 weeks).
  The VHI is a score formed by 5 parameters (vaginal elasticity, vaginal secretions, pH, epithelial mucous membrane, vaginal hydration). The final score defines the degree of atrophy in the genitourinary tract by assigning a single score to each parameter. The maximum possible score is 25, while the minimum possible score is 5.
The absolute change in Visual Analogous Scale (VAS). | From baseline to Day 30 (4 weeks) and Day 60 (up to 8 weeks).
  The absolute change in VAS, ranged between 0 (no pain) and 10 (worst possible pain), judged by the Principal Investigator.
The absolute change in Visual Analogous Scale (VAS) | From Day 0 to Day 30 (4 weeks) and Day 60 (up to 8 weeks).
  The absolute change in VAS ranged between 0 (no pain) and 10 (worst possible pain), judged by the subject.
The change of the Female Sexual Function Index (FSFI) score. | From Day 0 to Day 30 and Day 60 (up to 4 weeks and 8 weeks respectively).
  The FSFI is a validated questionnaire to measure the sexual functioning of women. The score ranges between 2 (minimum) and 36 (maximum).
Subject satisfaction evaluated by the Global Impression of Improvement (PGI-I) questionnaire | From Day 30 (4 weeks) to Day 60 (up to 8 weeks).
  The PGI-I is a transition single question scale, asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (Very much better) to 7 (Very much worse)
The change if the Nugent Score | From baseline to Day 60 (up to 8 weeks).
  The Nugent Score is a Gram stain scoring system for vaginal swabs to diagnose bacterial vaginosis, relying on scoring of individual types of organisms; a score of 0 to 10 is derived from a weighted combination of the following: large Gram-positive rods (lactobacilli; decrease in Lactobacillus scored as 0 to 4), small Gram-negative or Gram-variable rods (G. vaginalis or other anaerobes; scored as 0 to 4), and curved Gram-negative or Gram-variable rods (Mobiluncus spp.; scored as 0 to 2).
Viganal biopsy (optional) | From Day 0 up to Day 60 (up to 8 weeks).
  Evaluation of the mitotic activity of the mucosa (Ki-67 proliferation marker - %).
Participant's Questionnaire | From Day 0 to Day 30 and Day 60 (up to week 4 and 8 respectively).
  To register the overall discomfort and satisfaction of the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Ramus, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No